CLINICAL TRIAL: NCT00742118
Title: Effects of the Soluble Mediators of Mastocytes on the Intestinal Epithelial Barrier and of the entérique Nervous System During the Syndrome of the Irritable Bowel
Brief Title: Effects of the Soluble Mediators of Mastocytes on the Intestinal Epithelial Barrier and of the Enteric Nervous System During the Syndrome of the Irritable Bowel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Fondation de l'Avenir (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 05-API-08
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 (Experimental): patient with chronic inflammatory intestinal disease
  Interventions: Procedure: Colic biopsies
- 3 (Other): patient having no symptoms
  Interventions: Procedure: Colic biopsies
- 1 (Experimental): patient with irritable bowel syndrome
  Interventions: Procedure: Colic biopsies

INTERVENTIONS:
Procedure: Colic biopsies — colic biopsies and analysis
  Other Names: endoscopic biopsy

SUMMARY:
Patients with irritable bowel syndrome (IBS) have increased intestinal permeability. In addition, mucosal soluble mediators are involved in the pathophysiology of pain in IBS. The investigators aimed to investigate:

1. paracellular permeability in colonic biopsies of IBS patient
2. the ability of soluble factors from colonic biopsies to reproduce in vitro these alterations

ELIGIBILITY:
Inclusion Criteria:

* Patients needing coloscopy

Exclusion Criteria:

* Disrupted coagulation results
* Cancer even healed
* Known food allergy.
* Alcohol consumption >30g/day

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Para-cellular permeability | at time=0
Gap junction protein expression | at time=0
Inflammation molecule expression | at time=0
Digestive discomfort degree | at time=0

CONTACTS AND LOCATIONS:
Overall Officials: Thierry PICHE, PhD, Principal Investigator — Department of Gastroenterology
Locations (1):
- Department of gastroenterology, Hopital Archet 2, Nice, France